CLINICAL TRIAL: NCT00302432
Title: The Effect of Cigarette Holders, Plastic Menthol Cigarettes, and Cognitive Behavioral Therapy for Smoking Reduction Among Schizophrenia Inpatients: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lev-Hasharon Mental Healtlh Center (Other Government)
Responsible Party: Dr. Rudinski, Lev Hasharon Mental Health Center
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: LH16/2005.CTIL
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Schizophrenia; Heavy Smoking
Keywords: smoking reduction; group therapy; cigarette holders; "Flowers Menthol"
MeSH Terms: conditions — Schizophrenia; Smoking Reduction | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior therapy, cigarette holders, Flowers Menthol

SUMMARY:
This study aims:

1. to assess the effect of smoking reduction programs (behavior therapy alone or behavior therapy with cigarette holders; "Flowers Menthol" plastic cigarettes with menthol) on cigarette smoking habits in an antipsychotic treated schizophrenia population.

DETAILED DESCRIPTION:
Smoking is a leading preventable cause of death in the western world. The highest incidence of smoking is among psychiatric inpatients. The issue of smoking among psychiatric patients needs to be addressed, since this population already suffers from physical comorbidity and reduced life expectancy (Brown et al., 2000), which increase with smoking, considering the additional risk factors for cardiovascular diseases: obesity, high cholesterol, diabetes. In addition the increased risk factors associated with second generation antipsychotic treatment need to be considered. Significant financial expenditures for the purchase of cigarettes, from an already extremely limited budget (Steinberg et al., 2004) should be taken into account. Psychiatric patients who smoke spend up to 30% of their welfare payments on cigarettes.

A survey performed in our mental health center revealed that over 30% of the patients who smoke are interested in specific treatment to reduce/stop smoking (Melamed et al., unpublished). Our survey found that The expressed desire of the patients to quit smoking and the known dangers of smoking, especially in this population, reflect the importance of integrating smoking reduction/cessation programs into the treatment regimens of psychiatric inpatients.

Treatment options to promote smoking cessation include hypnosis (Spiegel et la., 1993; Weizman et al., 2004), behavior therapy (Addington et al., 1998), group therapy (Addington, 1998), nicotine replacement therapies (NRT) (Fant et al., 2000), and pharmacotherapy such as bupropion (George et al., 2002).

Since it is recommended that many smoking cessation treatment options such as NRT (nicotine transdermal patches or nicotine polacrilex gum, nasal spray, cigarette filters and nicotine inhalers) should not be used together with actual nicotine intake we decided to gradually introduce the issue of smoking reduction/cessation to the inpatient population, by initially introducing a program for smoking reduction.

Smoking reduction options include:

1. Cigarette holders
2. "Flowers Menthol"
3. Behavior therapy, including various relaxation techniques

Methods Study population: 60 subjects will be drawn from the inpatient population of Lev-Hasharon Mental Health Center, and divided into 4 groups of 15 participants each.

Inclusion criteria

1. Age 18-65 male or female.
2. DSM -IV criteria for chronic schizophrenia or schizoaffective disorder.
3. Ability and willingness to sign informed consent for participation in the study.
4. Patients' expressed interest in participating in a smoking-reduction program
5. Smoking a minimum of 20 cigarettes daily, for 6 months prior to the study period, as per patient report.
6. Patients treated with antipsychotic agents. Exclusion criteria

1- Significant physical illness. 2- Evidence of organic brain damage , mental retardation , alcohol or drug abuse.

3- Contraindication to amantadine treatment. 4- Pregnant or nursing female patients.

Duration of study will be 6 weeks. Patients will be assigned to one of 4 the intervention groups. Group assignment will be according to the department where the patient is hospitalized.

Group 1 - Behavior therapy only Group 2 - Behavior therapy with cigarette holders Group 3 - Behavior therapy with "Flowers Menthol" There will be no restrictions regarding the type of antipsychotic medication (typical or atypical) that participants are currently treated with.

Proposed study duration is 6 weeks. All patients will participate in 5 weekly behavioral group therapy sessions for smoking reduction. Each department will have a staff member devoted to smoking reduction "smoking supervisors" , who will accompany the patients throughout the week, advising, counseling, and supporting during crises.

Group 1 will have behavioral group therapy for smoking reduction, with not additional intervention.

Group 2 will be administered plastic cigarette holders. The nursing staff will distribute the holders one at a time. Used holders will be returned to the "smoking supervisor" when the sieve is blocked (usually after five cigarettes).

Group 3 will be administered Flowers Menthol (smokeless inhalers), one per day, by the "smoking supervisor". Used devices will be returned to him/her.

After receiving a detailed explanation of study procedures patients will sign informed consent. Throughout the study period, cigarettes will be distributed freely. Participants will fill out tables recording the number of cigarettes smoked, with the help of their "smoking supervisors".

Instruments

Patients will be assessed at baseline, and end of week 6 with the following instruments:

Clinical Rating Scales The patients' mental condition will be assessed with the Positive and Negative Syndrome Scale (PANSS) (Kay et al, 1987), Clinical Global Impression (CGI) scale for psychosis (Guy,1976), Hamilton Rating Scale for Depression (HAM-D) (Hamilton,1960), Simpson Angus Scale for extrapyramidal side effects (SAS) (Simpson and Angus 1970). Assessment of smoking dependence The Fagerstrom Tolerance Questionnaire for Nicotine Dependence (FTND Fagerstrom KO 1978) is useful and simple to administer for the evaluation of nicotine dependence.

Weekly table for self-report of the number of cigarettes smoked will be filled out by participants with the help of the "smoking supervisors".

Subjective Quality of Life Quality of life enjoyment and satisfaction questionnaire -abbreviated version (Q-LES-Q-18) (Ritsner et al., 2005).

Statistical analysis Appropriate statistical analysis will be performed including ANOVA with repeated measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 male or female.
2. DSM -IV criteria for chronic schizophrenia or schizoaffective disorder.
3. Ability and willingness to sign informed consent for participation in the study.
4. Patients' expressed interest in participating in a smoking-reduction program
5. Smoking a minimum of 20 cigarettes daily, for 6 months prior to the study period, as per patient report.
6. Patients treated with antipsychotic agents.

Exclusion Criteria:

1. Significant physical illness.
2. Evidence of organic brain damage , mental retardation , alcohol or drug abuse.
3. Pregnant or nursing female patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Assessment of smoking dependence: | 6 weeks
The Fagerstrom Tolerance Questionnaire for Nicotine Dependence (FTND) | 6 weeks
Weekly table for self-report of the number of cigarettes smoked will be filled out by participants with the help of the "smoking supervisors". | 6 weeks
Subjective Quality of Life: | 6 weeks
Quality of life enjoyment and satisfaction questionnaire -abbreviated version | 6 weeks

SECONDARY OUTCOMES:
Clinical Rating Scales: | 6 weeks
Positive and Negative Syndrome Scale (PANSS) | 6 weeks
Clinical Global Impression (CGI) scale for psychosis | 6 weeks
Hamilton Rating Scale for Depression (HAM-D) | 6 weeks
Simpson Angus Scale for extrapyramidal side effects (SAS) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Rudinski, MD, Principal Investigator — Lev-Hasharon MHC; Yuval Melamed, MD, MHA, Study Director — Lev-Hasharon MHC; Olga Preisman, MD, Study Chair — Lev-Hasharon MHC; Deby Peres, MD, Study Chair — Lev-Hasharon.MHC; Marc Gelkopf, Phd, Study Chair — Lev-Hasharon MHC; Sigalit Noam, RN, BA, Study Chair — Lev-Hasharon MHC; Arturo Lerner, MD, Study Chair — Lev-Hasharon MHC; Avi Bleich, MD, MPH, Study Director — Lev-Hasharon MHC
Locations (1):
- Lev-Hasharon MHC, Netanya, Israel